CLINICAL TRIAL: NCT07385625
Title: The Study for Evaluation of Acute Phase Safety and Efficacy of 'Pivot Bridge' to Short-term Treat Functional Tricuspid Regurgitation
Brief Title: Acute Safety and Efficacy of the Pivot Bridge System for Functional Tricuspid Regurgitation
Acronym: Pivot TR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tau-MEDICAL Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCP-IT2-08
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Tricuspid Regurgitation Functional
Keywords: Tricuspid Regurgitation; SPACER; Pivot Bridge
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: This study uses a self-controlled case series design in which each participant serves as their own control, with the period of prior medical therapy (Medical Treatment, MT) defined as the control period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients ≥18 Years With Massive or Greater Functional Tricuspid Regurgitation on Medical Therapy (Experimental): Patients aged 18 years or older with massive or greater functional tricuspid regurgitation who have received medical therapy (diuretics and/or pharmacological treatment) for at least 1 month
  Interventions: Device: Pivot Bridge

INTERVENTIONS:
Device: Pivot Bridge — The investigational "Pivot Bridge" device will be inserted through a small incision in the femoral vein and guided to the heart using a catheter. The Pivot Bridge device is designed to sit in the space where the valve isn't closing, helping the flaps of the valve to close tightly and reducing the amount of blood leaking back through the valve.

SUMMARY:
The purpose of this clinical trial is as follows.

To assess the safety of the investigational medical device "Pivot Bridge" in participants aged 18 years or older with massive or greater functinal tricuspid regurgitation (TR) who have received medical therapy (diuretics/pharmacological treatment) for at least one month.

To evaluate clinical outcomes related to improvement of tricuspid regurgitation symptoms following implantation of the "Pivot Bridge" device, including procedure success and clinical success.

This study is designed as a self-controlled case series without a separate control group. The participant's non-exposure period to the investigational medical device, consisting of prior medical therapy (Medical Treatment, MT), is defined as the control period. The study compares (1) a period of fixed-dose medical therapy maintained for up to one week prior to application of the investigational medical device, and (2) a period during which the investigational medical device is temporarily implanted (within 1 week) in conjunction with medical therapy (Pivot Bridge, PB).

To quantitatively evaluate the efficacy of the investigational medical device in inducing improvement of tricuspid regurgitation, the following are assessed:

1. improvement in regurgitation severity from baseline to Day 4-7 during fixed-dose medical therapy (ΔMT), and
2. improvement from pre-application to the time of device removal following additional application of the Pivot Bridge (ΔPB).

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria will be enrolled

* Adults aged 18 years or older at the time of screening
* Subjects who have received appropriate medical treatment (diuretics/medical therapy) for tricuspid regurgitation for at least 1 month prior to participation in this clinical trial
* Subjects who, at the screening visit, are assessed by transthoracic echocardiography (TTE) to have functional tricuspid regurgitation severity of Massive (4+) or greater, as defined by Tricuspid Valve Academic Research Consortium classification, and who have clinical symptoms corresponding to New York Heart Association (NYHA) functional class II or higher
* Subjects who, at the screening visit, are found on TTE or cardiac computed tomography (CT) to have a right ventricle (RV) larger than the left ventricle (LV)
* Subjects who, at the screening visit, are found on cardiac CT to have an annular diameter of 40 mm or greater
* Subjects for whom the Heart Team, consisting of at least one cardiologist (specialist in cardiology) and at least one cardiac surgeon, has determined that surgical treatment for isolated Tricuspid Regurgitation is required
* Subjects who voluntarily decide to participate in this clinical trial and provide written informed consent on the subject consent form
* Subjects who are able to understand and comply with the investigator's instructions and participate throughout the entire clinical trial period

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded

* Subjects in whom thrombus or embolic material is identified on echocardiography or cardiac computed tomography (CT) performed at the screening visit
* Subjects who have uncorrected coagulation disorders as shown by clinical laboratory tests performed at the screening visit
* Subjects who cannot use anticoagulant agents
* Subjects who, prior to participation in this clinical trial, have experienced major bleeding due to the use of anticoagulants (minor bleeding such as controllable epistaxis does not apply) requiring treatment, or who have had severe anemia necessitating hospitalization
* Subjects who, prior to participation in this clinical trial, have had devices such as an implantable cardioverter defibrillator (ICD) or a pacemaker implanted
* Subjects who, based on echocardiography and cardiac CT performed at the screening visit, are judged by the investigator to have anatomical structures unsuitable for implantation of the investigational medical device
* Subjects who, based on clinical laboratory tests performed at the screening visit, have a platelet count of ≤80,000/µL
* Subjects who, based on echocardiography performed at the screening visit, have pulmonary hypertension with TR Vmax ≥3.5 m/s
* Subjects who, based on echocardiography performed at the screening visit, have left ventricular ejection fraction (LVEF) <50%
* Subjects who, within 3 months prior to participation in this clinical trial, have had active gastrointestinal bleeding or have undergone gastrointestinal procedures (subjects with a risk of gastrointestinal bleeding)
* Subjects who, within 30 days prior to participation in this clinical trial, have a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA)
* Subjects who, within 30 days prior to participation in this clinical trial, have a history of myocardial infarction (MI)
* Subjects with active infective endocarditis requiring antibiotic therapy
* Subjects with severe terminal illnesses (e.g., malignant tumors, end-stage pulmonary disease, end-stage liver disease, end-stage renal failure)
* Subjects who, based on echocardiography performed at the screening visit, have moderate or severe aortic, pulmonary, or mitral stenosis
* Subjects who, based on echocardiography performed at the screening visit, are found to have calcification of the tricuspid valve leaflets that would affect the procedure
* Subjects who, based on echocardiography performed at the screening visit, are found to have masses, thrombi, or proliferative lesions in the right heart system, femoral vein, or inferior vena cava
* Subjects who, within 30 days prior to participation in this clinical trial, have participated in another clinical trial
* Pregnant or lactating women, and women planning to become pregnant during the study period
* Women of childbearing potential who are not using medically acceptable methods of contraception
* Subjects who, in addition to the above, are deemed by the investigator to have clinically significant findings that make them inappropriate for participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Procedure Success Based on Improvement in Tricuspid Regurgitation Severity | Visit 2 (Baseline, MT Day 0), Visit 3 (MT Day 4-7), Visit 3 (PB Day 4-7)
  Proportion of subjects achieving at least a 1-grade improvement in tricuspid regurgitation (TR grade) according to Tricuspid Valve Academic Research Consortium definitions

SECONDARY OUTCOMES:
Clinical Success Based on Clinical Improvement | Visit 2 (Baseline, MT Day 0), Visit 3 (MT Day 4-7), Visit 3 (PB Day 4-7)
  The number of participants who experienced at least 1 drop in their TR grade from Baseline
Clinical Success Based on Clinical Improvement(1) | Visit 2 (Baseline, MT Day 0), Visit 3 (MT Day 4-7), Visit 3 (PB Day 4-7)
  Changes in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) score (a measure of symptoms, physical limitation, social limitations and quality of life domains) from baseline. Participants will be asked to tick a box on a scale indicating how each domain affects their life (e.g. scales range from extremely limited to not at all limited, from every morning/night to never over the past 2 weeks, from completely dissatisfied to completely satisfied). The responses will be used to calculate an average score on a scale of 0 to 100. A higher score equates to better outcomes (i.e. fewer symptoms, better physical and social function, improved quality of life).
Clinical Success Based on Clinical Improvement(2) | Visit 2 (Baseline, MT Day 0), Visit 3 (MT Day 4-7), Visit 3 (PB Day 4-7)
  Changes in eGFR (estimated glomerular filtration rate) from baseline
Clinical Success Based on Clinical Improvement(3) | Visit 2 (Baseline, MT Day 0), Visit 3 (MT Day 4-7), Visit 3 (PB Day 4-7)
  Number of participants with at least 1 level of improvement in pitting edema from baseline
Clinical Success Based on Clinical Improvement(4) | Visit 2 (Baseline, MT Day 0), Visit 3 (MT Day 4-7), Visit 3 (PB Day 4-7)
  Number of participants with improvement in New York Heart Association (NYHA) functional class (system to classify the severity of heart failure symptoms) from baseline
Clinical Success Based on Clinical Improvement(5) | Visit 2 (Baseline, MT Day 0), Visit 3 (MT Day 4-7), Visit 3 (PB Day 4-7)
  Changes in echocardiogram (measurements and assessments of the heart's structure and function) as assessed by the central "Core Lab" reader
Clinical Success Based on Anatomical Improvement | Visit1 (Screening), Visit 3 (PB Day 4-7)
  Anatomical improvement : right ventricular volume, tricuspid valve annulus area, and other CT core lab analysis parameters
Clinical Success Within 3 Days After Device Removal | Visit 2 (Baseline, MT Day 0), Visit 3 (Post-removal)
  Changes in echocardiogram (measurements and assessments of the heart's structure and function) as assessed by the central "Core Lab" reader
Clinical Success at 1 Month After Device Removal | Visit 2 (Baseline, MT Day 0), Visit 4 (End of Study Visit, PB+ 1 Month)
  Changes in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) score (a measure of symptoms, physical limitation, social limitations and quality of life domains) from baseline. Participants will be asked to tick a box on a scale indicating how each domain affects their life (e.g. scales range from extremely limited to not at all limited, from every morning/night to never over the past 2 weeks, from completely dissatisfied to completely satisfied). The responses will be used to calculate an average score on a scale of 0 to 100. A higher score equates to better outcomes (i.e. fewer symptoms, better physical and social function, improved quality of life).
Clinical Success at 1 Month After Device Removal(1) | Visit 2 (Baseline, MT Day 0), Visit 4 (End of Study Visit, PB+ 1 Month)
  Changes in eGFR (estimated glomerular filtration rate) from baseline
Clinical Success at 1 Month After Device Removal(2) | Visit 2 (Baseline, MT Day 0), Visit 4 (End of Study Visit, PB+ 1 Month)
  Number of participants with at least 1 level of improvement in pitting edema from baseline
Clinical Success at 1 Month After Device Removal(3) | Visit 2 (Baseline, MT Day 0), Visit 4 (End of Study Visit, PB+ 1 Month)
  Number of participants with improvement in New York Heart Association (NYHA) functional class (system to classify the severity of heart failure symptoms) from baseline
Clinical Success at 1 Month After Device Removal(4) | Visit 2 (Baseline, MT Day 0), Visit 4 (End of Study Visit, PB+ 1 Month)
  Changes in echocardiogram (measurements and assessments of the heart's structure and function) as assessed by the central "Core Lab" reader

CONTACTS AND LOCATIONS:
Overall Officials: Geu-Ru Hong, MD, PhD, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (4):
- South Korea (4):
  - Keimyung University Dongsan Hospital, Daegu, Dalseo-gu
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Yonsei University Health System, Severance Hospital, Seoul, Seodaemun-gu
  - Asan Medical Center, Seoul, Songpa-gu

IPD SHARING:
Plan to Share IPD: No